CLINICAL TRIAL: NCT04261907
Title: A Randomized, Open-label, Multi-centre Clinical Trial Evaluating and Comparing the Safety and Efficiency of ASC09/Ritonavir and Lopinavir/Ritonavir for Confirmed Cases of Pneumonia Caused by Novel Coronavirus Infection
Brief Title: Evaluating and Comparing the Safety and Efficiency of ASC09/Ritonavir and Lopinavir/Ritonavir for Novel Coronavirus Infection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There were no more subjects enrolled.
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASC09F-CTP-ZY-01
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2020-02

CONDITIONS: 2019-nCoV
MeSH Terms: interventions — TMC-310911; Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASC09/ritonavir group (Experimental): ASC09/ritonavir (300mg/100mg tablet)+conventional standardized treatment
  Interventions: Drug: ASC09/ritonavir group
- lopinavir/ritonavir group (Active Comparator): Lopinavir/ritonavir tablet (200mg / 50mg tablet)+conventional standardized treatment
  Interventions: Drug: lopinavir/ritonavir group

INTERVENTIONS:
Drug: ASC09/ritonavir group — ASC09/ritonavir(300mg/100mg tablet), one tablet each time, twice daily, for 14 days, +conventional standardized treatment
  Arms: ASC09/ritonavir group
Drug: lopinavir/ritonavir group — Lopinavir/ritonavir tablets(200mg / 50mg tablet), two tablets each time, twice daily, for 14 days, +conventional standardized treatment
  Arms: lopinavir/ritonavir group

SUMMARY:
Base on Arbidol antiviral therapy,the investigators conduct a randomized, open-label trial to evaluate and compare the safety and efficacy of ASC09 /ritonavir and lopinavir/ritonavir in patients with 2019-nCoV pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged between 18 and 75 years, extremes included, male or female
* 2. Laboratory (RT-PCR) and clinical symptoms confirmed case of 2019-nCoV pneumonia, according to the official guideline "Pneumonia Diagnosis and Treatment Scheme for Novel Coronavirus Infection (Trial Version 5)"
* 3. Hospitalised with a new onset respiratory illness (≤7 days since illness onset)
* 4. No family planning within six months, and agree to take effective contraceptive measures throughout the study and for at least 30 days after the final study drug dose
* 5. Must agree not to enroll in another study of an investigational agent prior to completion of Day 30 of study
* 6. Informed Consent Form (ICF) signed voluntarily

Exclusion Criteria:

* 1. Severe 2019-nCoV pneumonia met one of the following criteria: respiratory distress, RR ≥ 30 times / min, or SaO2 / SpO2 ≤ 93% in resting state, or arterial partial pressure of oxygen (PaO2) /concentration of oxygen (FiO2) ≤ 300mmHg (1mmHg = 0.133kpa)
* 2. Critical severe 2019-nCoV pneumonia met one of the following criteria: respiratory failure and mechanical ventilation required, or shock, or combined with other organ failure required ICU monitoring treatment
* 3. Severe liver disease (e.g. Child Pugh score ≥ C, AST > 5 times upper limit)
* 4. Known allergic reaction to any of components of ASC09 / ritonavir compound tablets
* 5. Patients with definite contraindications in the label of ritonavir
* 6. Positive serum pregnancy test result for women with childbearing potential at screening
* 7. Using HIV protease inhibitor drugs
* 8. Not suitable for the study, in the opinion of the Investigator (e.g. patient may be transferred to another hospital during the study period, patient with multiple basic diseases, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
The incidence of composite adverse outcome | 14 days
  Defined as(one of them) SPO2≤ 93% without oxygen supplementation, PaO2/FiO2 ≤ 300mmHg or RR ≥ 30 breaths per.

SECONDARY OUTCOMES:
Time to recovery | 14 days
  Clinical recovery was defined as( one of them): sustained (48 hours) alleviation of illness based on symptom scores (fever, cough,diarrhea, myalgia, dyspnea) all being absent and no evidence for progression (newly-presented dyspnea, SpO2 decline ≥3%, respiratory rate ≥ 24 breaths per min without supplemental oxygen). Or undectable viral RNA.
Rate of no fever | 14 days
Rate of no cough | 14 days
Rate of no dyspnea | 14 days
Rate of no requring supplemental oxygen | 14 days
Rate of undectable viral RNA | 14 days
Rate of mechanical ventilation | 14 days
Rate of ICU admission | 14 days
Time and rate of laboratory indicators related to disease improvement to return to normal | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Yunqing Qiu, Master, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The first affiliated hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang Province, P.R. China, China

IPD SHARING:
Plan to Share IPD: No